CLINICAL TRIAL: NCT04186650
Title: Phase I/II ex Vivo Gene Therapy Clinical Trial for RDEB Using Autologous Skin Equivalent Grafts Genetically Corrected With a COL7A1-encoding SIN Retroviral Vector
Brief Title: Ex Vivo Gene Therapy Clinical Trial for RDEB Using Genetically Corrected Autologous Skin Equivalent Grafts
Acronym: EBGraft
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C12-48; 2016-002790-35 (EudraCT Number)
Record Dates: First submitted 2019-11-25; First posted 2019-12-05 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Epidermolysis Bullosa Dystrophica, Recessive
Keywords: Genetic Therapy; Autologous Skin Graft; SIN retroviral vector; Type VII collagen; COL7A1
MeSH Terms: conditions — Epidermolysis Bullosa Dystrophica

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Autologous genetically modified tissue-engineered skin graft (Experimental): Graft of SIN RV-mediated COL7A1 gene-modified autologous skin equivalent
  Interventions: Biological: COL7A1-SIN retroviral vector engineered autologous tissue-engineered skin

INTERVENTIONS:
Biological: COL7A1-SIN retroviral vector engineered autologous tissue-engineered skin — Graft of SIN RV-mediated COL7A1 gene-modified autologous skin equivalent

SUMMARY:
This phase I/II clinical trial aims to treat 3 adult subjects with Recessive Dystrophic Epidermolysis Bullosa, expressing residual C7 levels, by genetically corrected autologous skin equivalent grafts on selected areas (up to 300 cm2).

DETAILED DESCRIPTION:
Recessive Dystrophic Epidermolysis Bullosa (RDEB) is a severe orphan genetic disease responsible for skin and mucosal detachments due to a loss of adhesion of the epidermis to the underlying dermis. The disease is caused by loss of function mutations of the COL7A1 encoding type VII collagen (C7) which forms anchoring fibers, which are essential structures for dermal-epidermal adherence. Current treatments are only symptomatic and do not effectively treat or prevent the occurrence of cutaneous and mucosal detachments responsible for local and systemic complications that threaten the vital prognosis.

EBGRAFT is a prospective open-label international monocentric phase I/II clinical trial. It aims to treat 3 adult subjects with RDEB, expressing residual C7 levels, by genetically corrected autologous skin equivalent grafts.

The skin equivalent consists of keratinocytes and fibroblasts from the patient, genetically corrected ex vivo with a secure Self INactivating (SIN) retroviral vector expressing the COL7A1 cDNA under the control of the ubiquitous human promoter EF1a.

Each patient will be grafted sequentially at Necker Hospital in Paris using autologous genetically corrected skin equivalents of approximately 300 cm2 (up to 6 grafts of 50 cm2 each).

The main objective is to evaluate the safety of autologous skin equivalent grafts genetically corrected with a SIN COL7A1 retroviral vector (RV) in adults with RDEB.

The secondary objectives are:

1. To evaluate the efficacy of transplanting autologous skin equivalent genetically corrected with RV SIN COL7A1 in adults with RDEB.
2. To evaluate the immune response against recombinant type VII collagen (C7).

This clinical trial should evaluate whether the grafting of these genetically corrected autologous skin equivalents is well tolerated and whether they restore normal dermal-epidermal adherence of the grafted areas. The proposed treatment aims to obtain a permanent correction of the grafted areas, allowing skin healing and reducing pain. It has the potential to reduce itching, to prevent the occurrence of blisters and skin detachments, reduce the risk of infections, the duration and cost of care and also the risk of development of squamous cell carcinomas in the grafted areas.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical and molecular diagnosis of RDEB with confirmed bi-allelic COL7A1 mutations
2. Reduced staining of C7 on skin biopsy, measured by immunofluorescence microscopy (IF)
3. A reduced number of/or morphologically abnormal anchoring fibrils confirmed by TEM
4. Detection of non-collagenous-1 domain (NC-1) of C7 on skin biopsy, measured by immunofluorescence microscopy (IF) and/or Western blot (WB) analysis
5. Presence of ≥100cm2 of blistered and/or erosive skin areas including chronic wounds suitable for skin grafting
6. Ability to undergo anaesthesia for skin grafting procedures
7. Subjects aged 18 years, willing and able to give informed consent

Exclusion Criteria:

1. Recipients of other investigational medicinal products within 6 months prior to enrolment into this study
2. Past medical history of biopsy proven skin malignancy
3. Immunotherapy including oral corticosteroids (Prednisolone >1mg/kg) for more than one week (intranasal and topical preparations are permitted) or chemotherapy within 60 days of enrolment into this study
4. Known allergy to any of the constituents of the investigational medicinal product (IMP) including Penicillin
5. Subjects with BOTH:

   * positive serum antibodies to C7 confirmed by ELISA and
   * positive IIF with binding to the base of salt split skin and/or
   * positive Western blot
6. Positive results for HIV, Hepatitis BsAg, Hepatitis BcAb, Hepatitis C IgG, HTLV1&2 or Syphilis serology
7. Clinically significant medical, psychological or laboratory abnormalities limiting the ability of the subject to travel to the trial site(s) and to undergo grafting and follow-up procedures, as determined by the Investigator
8. Absence of adequate social support
9. Subjects who are pregnant, breast-feeding or of child-bearing potential who are neither abstinent nor practicing an acceptable means of contraception when this is in line with the usual and preferred lifestyle of the subject, as determined by the Investigator, for the duration of the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2020-01-10 (Actual); Primary Completion 2027-06-09 (Estimated); Study Completion 2027-06-09 (Estimated)

PRIMARY OUTCOMES:
Safety of grafting SIN RV-mediated COL7A1 gene-modified autologous skin equivalent: Adverse Events (AE), Serious Adverse Events (SAEs), Adverse Reactions (ARs) and Serious Adverse Reactions (SARs) | Month 12 post grafting.
  The primary objective is to evaluate the safety of autologous autologous skin equivalent grafts genetically corrected with a SIN COL7A1 retroviral vector (RV) in adults with RDEB
  Primary Endpoints:
  Record of Adverse Events (AE), Serious Adverse Events (SAEs), Adverse Reactions (ARs) and Serious Adverse Reactions (SARs).

SECONDARY OUTCOMES:
Change in C7 protein expression | Month 1, Month 3, Month 6, Month 12 post grafting.
  Skin biopsy analysis of grafted skin compared to baseline for :
  C7 protein expression by immunofluorescence microscopy (IF) using several specific antibodies
Change in anchoring fibrils number | Month 1, Month 3, Month 6, Month 12 post grafting.
  Count of anchoring fibril (AF) at the dermal-epidermal junction (DEJ) by transmission electron microscopy (TEM) will be performed on skin biopsies and
Change in scar quality: Vancouver Scar Scale (VSS) | Month 1, Month 2, Month 3, Month 6, Month 12 post grafting.
  Scar quality will be measured using the Vancouver Scar Scale (VSS) and compared to baseline at several time points. Minimum value=0, Maximum value=12. Lower value is better.
Changes in blister number over the grafted skin | Month 1, Month 2, Month 3, Month 6, Month 12 post grafting.
  Blister formation will be monitored and counted by a skilled dermatologist and compared to baseline at several time points.
Changes in clinical appearance of grafted skin | Month 1, Month 2, Month 3, Month 6, Month 12 post grafting.
  Clinical appearance of the grafted skin areas will be assessed by 3D photographic reconstruction using a CANFIELD Vectra H1 device and compared to baseline at several time points.
Changes in pruritus of grafted skin | Month 1, Month 2, Month 3, Month 6, Month 12 post grafting.
  Pruritus will be measured by the 5D pruritus score and compared to baseline at several time points. Minimum value=4, Maximum value=35. Lower value is better.
Change in Quality of life: QOLEB questionnaire (Quality of Life for Epidermolysis Bullosa) | Month 1, Month 2, Month 3, Month 6, Month 12 post grafting.
  Quality of life will be measured using the specific QOLEB questionnaire (Quality of Life for Epidermolysis Bullosa) and compared to baseline at several time points.
  Minimum value=0, Maximum value=51. Lower value is better.
Change in Birmingham Epidermolysis Score (BEBS) | Month 1, Month 2, Month 3, Month 6, Month 12 post grafting.
  Change in disease severity will be assessed by the Birmingham Epidermolysis Score (BEBS).
  Score will be compared to baseline at several timepoints. Minimum value=0, Maximum value=100. Lower value is better.
Change in Epidermolysis Bullosa Disease Activity and Scarring Index (EBDASI) - Activity | Month 1, Month 2, Month 3, Month 6, Month 12 post grafting.
  Change in disease severity will be assessed by the Epidermolysis Bullosa Disease Activity and Scarring Index (EBDASI). Score will be compared to baseline at several timepoints. Score measure activity (minimum value=0, maximum value=276). Lower value is better.
Change in Epidermolysis Bullosa Disease Activity and Scarring Index (EBDASI) - Damage | Month 1, Month 2, Month 3, Month 6, Month 12 post grafting.
  Change in disease severity will be assessed by the Epidermolysis Bullosa Disease Activity and Scarring Index (EBDASI). Score will be compared to baseline at several timepoints. Score measure damage (minimum value=0, maximum value=230). Lower value is better.
Change in instrument for Scoring Clinical Outcomes of Research for Epidermolysis Bullosa (iscorEB). | Month 1, Month 2, Month 3, Month 6, Month 12 post grafting.
  Change in disease severity will be assessed by the instrument for Scoring Clinical Outcomes of Research for Epidermolysis Bullosa (iscorEB). Score will be compared to baseline at several timepoints. Minimum value=0, Maximum value=120. Lower value is better.
Evaluation of the humoral immune response against recombinant C7 | Month 1, Month 6, Month 12 post grafting.
  Detection of circulating anti-C7 antibodies in patient blood by ELISA and/or indirect immunofluorescence (IIF) on split skin at several time points
Evaluation of the cytotoxic immune response against recombinant C7 | Month 1, Month 6, Month 12 post grafting.
  Detection of T-cell responses to the full length C7 in patient blood by ELISPOT assay.

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Imagine Necker Hospital, Paris, France

REFERENCES:
- [Background] Gaucher S, Lwin SM, Titeux M, Abdul-Wahab A, Pironon N, Izmiryan A, Miskinyte S, Ganier C, Duchatelet S, Mellerio JE, Bourrat E, McGrath JA, Hovnanian A. EBGene trial: patient preselection outcomes for the European GENEGRAFT ex vivo phase I/II gene therapy trial for recessive dystrophic epidermolysis bullosa. Br J Dermatol. 2020 Mar;182(3):794-797. doi: 10.1111/bjd.18559. Epub 2019 Nov 27. No abstract available. PMID 31557321
- [Background] Titeux M, Pendaries V, Zanta-Boussif MA, Decha A, Pironon N, Tonasso L, Mejia JE, Brice A, Danos O, Hovnanian A. SIN retroviral vectors expressing COL7A1 under human promoters for ex vivo gene therapy of recessive dystrophic epidermolysis bullosa. Mol Ther. 2010 Aug;18(8):1509-18. doi: 10.1038/mt.2010.91. Epub 2010 May 18. PMID 20485266
- [Background] Hennig K, Raasch L, Kolbe C, Weidner S, Leisegang M, Uckert W, Titeux M, Hovnanian A, Kuehlcke K, Loew R. HEK293-based production platform for gamma-retroviral (self-inactivating) vectors: application for safe and efficient transfer of COL7A1 cDNA. Hum Gene Ther Clin Dev. 2014 Dec;25(4):218-28. doi: 10.1089/humc.2014.083. PMID 25381930